CLINICAL TRIAL: NCT05323786
Title: Effect of Topical Anesthesia on Hemodynamics During Induction in Patients Undergoing Cardiac Surgery: a Randomized Controlled Study
Brief Title: Hemodynamic Effect of Topical Anesthesia During Induction in Patients Undergoing Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Lili Cao, Professor, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TACTICS-Ⅱ
Record Dates: First submitted 2022-04-02; First posted 2022-04-12 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Disease; Valvular Heart Disease; Arrythmia
Keywords: Topical anesthesia; Atomization inhalation; Cardiac surgery; Hemodynamics; Endotracheal intubation
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases; Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The combined topical anesthesia induction group (Experimental): Inhalation of aerosolized surface anesthesia with 10 ml 2% lidocaine would be administered with an atomizer for 15 minutes prior to intravenous anesthesia. After the intravenous induction, a catheter would be inserted to provide the subglottic anesthesia with 3ml 2% lidocaine.
  Interventions: Procedure: The combined topical anesthesia induction group
- The routine induction group (Placebo Comparator): Inhalation of 10 ml 0.9% normal saline would be administered with an atomizer for 15 minutes prior to intravenous anesthesia. After the intravenous induction, 3ml 0.9% normal saline would be administered into subglottic airway with a catheter.
  Interventions: Procedure: The routine induction group

INTERVENTIONS:
Procedure: The combined topical anesthesia induction group — Inhalation of aerosolized surface anesthesia with 10 ml 2% lidocaine would be administered with an atomizer for 15 minutes prior to intravenous anesthesia. After the intravenous induction, a catheter would be inserted to provide the subglottic anesthesia with 3ml 2% lidocaine.
  Arms: The combined topical anesthesia induction group
Procedure: The routine induction group — Inhalation of 10 ml 0.9% normal saline would be administered with an atomizer for 15 minutes prior to intravenous anesthesia. After the intravenous induction, 3ml 0.9% normal saline would be administered into subglottic airway with a catheter.
  Arms: The routine induction group

SUMMARY:
Patients scheduled for cardiac surgery are fragile. Hemodynamic fluctuation might be associated with adverse outcomes. Therefore, it is essential to keep hemodynamics stable during and after the induction period. Previous studies have shown that topical anesthesia can provide excellent superior supraglottic and subglottic local anesthetic effects and can significantly reduce the dosage of intravenous anesthetics. Therefore, we designed this study to explore whether the combination of topical anesthesia and intravenous anesthetics could decrease the stress response of endotracheal intubation and keep hemodynamics stable during and after the induction period.

DETAILED DESCRIPTION:
Patients scheduled for cardiac surgery are often accompanied by cardiac insufficiency. Hemodynamic fluctuation might lead to disastrous events. Therefore, it is essential to keep hemodynamics stable during and after the induction period. The routine anesthesia induction strategy for cardiac surgery is to decrease stress response during endotracheal intubation by using large doses of opioids. However, high doses of opioids often leads to persistent and recurrent hypotension in patients from the anesthesia induction period to the beginning of the surgery. Previous studies have shown that topical anesthesia can provide excellent superior supraglottic and subglottic local anesthetic effects and can significantly reduce the dosage of intravenous anesthetics. Therefore, we designed this study to explore whether the combination of topical anesthesia and intravenous anesthetics could decrease the stress response of endotracheal intubation and keep hemodynamics stable during and after the induction period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years and younger than 75 years;
2. Patients scheduled to accept elective cardiac surgery;
3. Patients of New York Heart Association (NYHA) Ⅱ～Ⅲ level grade ;
4. Patients signed the informed consent form for the clinical study.

Exclusion Criteria:

1. Patients cannot cooperate to topical anesthesia;
2. Patients who had left heart assist devices other than intra-aortic balloon counterpulsation before surgery;
3. Patients treated with Extracorporeal Membrane Oxygenation (ECMO) prior to surgery;
4. Patients with aortic dissection;
5. Patients with difficult airway;
6. Patients with high sensitivity and hypersensitivity to lidocaine;
7. Patients with atrioventricular block;
8. Patients who have participated in other clinical studies during the last 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-21 (Actual)

PRIMARY OUTCOMES:
The area under the curve of baseline blood pressure | From 3 minutes after endotracheal intubation(T1) to 15 minutes after endotracheal intubation(T2). T1 is defined as 3 minutes after endotracheal intubation. T2 is defined as 15 minutes after endotracheal intubation. It will take up to 1hour or 2hours.
  The area under the curve (AUC) of blood pressure below baseline mean arterial pressure within 3 minutes to 15 minutes after endotracheal intubation

SECONDARY OUTCOMES:
The area under the curve of baseline blood pressure | From from the beginning of the general anaesthesia induction(T1) to 3 minutes after endotracheal intubation(T2). T1 is when midazolam is administered. T2 is defined as 3 minutes after endotracheal intubation. It will take up to 1hour or 2hours.
  AUC above baseline MAP (MAP-time integral) and below baseline MAP (MAP-time integral)
The highest and lowest values of arterial blood pressure | From the beginning of the general anaesthesia induction(T1) to 15 minutes after endotracheal intubation(T2). T1 is when midazolam is administered. T2 is defined as 15 minutes after endotracheal intubation. It will take up to 1hour or 2hours.
  The highest and lowest values of arterial blood pressure (SBP, DBP, MAP)
The types of vasoactive drugs used. | From the beginning of the general anaesthesia induction(T1) to 15 minutes after endotracheal intubation(T2). T1 is when midazolam is administered. T2 is defined as 15 minutes after endotracheal intubation. It will take up to 1hour or 2hours.
  The types of vasoactive drugs used ,such as the use of norepinephrine and dopamine.
The frequency of vasoactive drugs used. | From the beginning of the general anaesthesia induction(T1) to 15 minutes after endotracheal intubation(T2). T1 is when midazolam is administered. T2 is defined as 15 minutes after endotracheal intubation. It will take up to 1hour or 2hours.
  The frequency of vasoactive drugs used ,such as the use of norepinephrine and dopamine.
The incidence of arrhythmias. | From the beginning of the general anaesthesia induction(T1) to 15 minutes after endotracheal intubation(T2). T1 is when midazolam is administered. T2 is defined as 15 minutes after endotracheal intubation. It will take up to 1hour or 2hours.
  The incidence of arrhythmias, such as atrioventricular block, atrial fibrillation, ventricular tachycardia and so on.
cardiac systolic function:Left Ventricular Ejection Fraction (LVEF) | Beginning of the general anaesthesia induction(T1) is when midazolam is administered. T2 is when central venous catheterization is finished. It will take up to 1hour or 2hours.
  Left ventricular ejection fraction，a parameter of left ventricular systolic function. left ventricular ejection fraction (LVEF) (﹪)= stroke output (SV)/ left ventricular end-diastolic volume (LEDV)×100﹪，will be evaluated before induction of anesthesia and after central venous catheterization.
cardiac diastolic function:E/E' (the ratio of E peak and E') or E/A :(the ratio of E peak and A peak) | Beginning of the general anaesthesia induction(T1) is when midazolam is administered. T2 is when central venous catheterization is finished. It will take up to 1hour or 2hours.
  E/A ratio, one of the main parameter for evaluating diastolic function, indicated normal diastolic function when E/A >1, and decreased diastolic function when E/A < 1.It will be evaluated before induction of anesthesia(T1) and after central venous catheterization(T2).
tricuspid annular plane systolic excursion(TAPSE) | Beginning of the general anaesthesia induction(T1) is when midazolam is administered. T2 is when central venous catheterization is finished. It will take up to 1hour or 2hours.
  Tricuspid annular plane systolic excursion is a reliable indicator of right ventricular systolic function.It represents the longitudinal function of the RV and it should be measured in the apical four-chamber projection using one-dimensional echocardiography (M-mode) at the peak excursion of the tricuspid annulus (expressed in millimeters) from the end of diastole to the end of systole.It will be evaluated before induction of anesthesia(T1) and after central venous catheterization(T2).
Respiratory variation in inferior vena cava diameter (DIVC) | Beginning of the general anaesthesia induction(T1) is when midazolam is administered. T2 is when central venous catheterization is finished. It will take up to 1hour or 2hours.
  Respiratory variation in inferior vena cava diameter (DIVC) is a measure of capacity load.DIVC=(Maximum diameter of inferior vena cava - minimum diameter of inferior vena cava) ÷ maximum diameter of inferior vena cava
The number of patients with postoperative hoarseness. | Three days after the surgery
  Hoarseness was classified as mild, moderate and severe according to the severity.
The number of patients with postoperative sore throat. | Three days after the surgery
  Sore throats can be evaluated using the Numeric Pain Scale (NRS) pain numerical score(0-10 score, 0: no pain, 10: worst imaginable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Meng Lv, doctor, Principal Investigator — Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University
Locations (1):
- Meng-Lv, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Du W, Lv M, Chen T, Sun X, Wang J, Zhang H, Wei C, Liu Y, Qiao C, Wang Y. The effect of topical airway anesthesia on hemodynamic profiles during the induction period in patients undergoing cardiac surgery: Study protocol for a randomized controlled trial. Front Cardiovasc Med. 2022 Oct 10;9:992534. doi: 10.3389/fcvm.2022.992534. eCollection 2022. PMID 36299870